CLINICAL TRIAL: NCT01695590
Title: Phase 1/2, Multi-center, Open Label, Dose Escalation, Safety, Efficacy and PK Study of PRLX 93936 Administered IV 3 Days a Week for 3 Weeks Followed by a 9 Day Rest Period in Patients With Relapsed or Relapsed/Refractory Multiple Myeloma
Brief Title: Safety, Efficacy and Pharmacokinetic Study of PRLX 93936 in Patients With Multiple Myeloma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Prolexys Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRLX93936-0002
Record Dates: First submitted 2012-09-18; First posted 2012-09-28 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-05

CONDITIONS: Multiple Myeloma
Keywords: Myeloma; PRLX93936
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PRLX 93936 (Experimental): PRLX 93936 administered IV 3 days a week (Monday, Wednesday and Friday) for 3 weeks followed by a 9 day rest period = 1 cycle
  Interventions: Drug: PRLX 93936

INTERVENTIONS:
Drug: PRLX 93936 — PRLX 93936 administered IV 3 days a week (Monday, Wednesday and Friday) for 3 weeks followed by a 9 day rest period = 1 cycle, multiple cycles may be administered

SUMMARY:
To determine the maximum tolerated dose of, and response to, PRLX 93936 as treatment for patients with relapsed or relapsed/refractory multiple myeloma.

DETAILED DESCRIPTION:
* To determine the maximum tolerated dose (MTD) and the dose limiting toxicities (DLT) of PRLX 93936 administered IV 3 days a week (Monday, Wednesday and Friday) for 3 weeks followed by a 9 day rest period, as treatment for patients with relapsed or relapsed/refractory multiple myeloma.
* To establish the dose of PRLX 93936 recommended for future studies.
* To characterize potential toxicities of PRLX 93936.
* To assess the pharmacokinetic profile of PRLX 93936.
* To evaluate response to treatment, time to response (TTR) and duration of response.
* To evaluate time to progression (TTP).

ELIGIBILITY:
Inclusion Criteria:

* Patient must have a diagnosis of multiple myeloma and have relapsed or relapsed/refractory disease.
* Patient must have received ≥ 2 prior anti-myeloma regimens including a proteasome inhibitor and/or immunomodulatory agent.
* Patient currently requires systemic therapy.
* Patient has measurable disease.
* Age ≥ 18 years
* Karnofsky performance status ≥ 60%
* ECOG performance 0, 1 or 2
* Life expectancy of at least three months
* Able to take acetaminophen
* Not pregnant
* Patient must have recovered from toxicities incurred as a result of any previous anti-myeloma therapy or recovered to baseline.
* Patients who received an autologous stem cell transplant must be ≥ 3 months post-transplant and all associated toxicities must have resolved to ≤ CTCAE Grade 1.
* QT intervals of QTc ≤ 500 msec

Exclusion Criteria:

* POEMS syndrome
* Plasma cell leukemia
* Primary amyloidosis
* Patient has smoldering multiple myeloma or monoclonal gammopathy of unknown significance (MGUS).
* Evidence of spinal cord compression or CNS complication unless controlled by appropriate therapy.
* Patient received chemotherapy or other anti-cancer therapy that may be active against multiple myeloma within 3 weeks prior to the first dose of PRLX 93936.
* Patient received nitrosureas within 6 weeks prior to the first dose.
* Patient received corticosteroids within 2 weeks prior to the first dose.
* Patient received plasmapheresis within 4 weeks prior to the first dose.
* Patient had major surgery within 4 weeks prior to the first dose.
* Patient had an allogeneic stem cell transplant within 6 months before first dose of PRLX 93936 or has evidence of graft versus host disease.
* Patient is taking any therapy concomitantly that may be active against multiple myeloma.
* Patient is currently receiving medication(s) that are principally metabolized via the cytochrome P450 3A4 enzyme pathway.
* Use of any investigational agents within 28 days or 5 half-lives (whichever is shorter) of study treatment.
* Patient has peripheral neuropathy of Grade 3 or greater intensity, or painful Grade 2, as defined by the NCI CTC.
* Patient had a myocardial infarction within 6 months of enrollment or has NYHA Class III or IV heart failure uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities.
* Abnormal LVEF (< LLN for the institution for a patient of that age) on echocardiogram
* Patient has poorly controlled hypertension, diabetes mellitus, or other serious medical or psychiatric illness that could potentially interfere with the completion of treatment according to protocol.
* Patient had a malignancy other than multiple myeloma within 3 years before enrollment, with the exception of adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, in situ breast cancer, or in situ prostate cancer.
* Patient's clinical laboratory values meet any of the following criteria within the 7 days prior to Study Day 1:

  * Bilirubin > 1.5 times ULN
  * AST (SGOT), ALT (SGPT) and Alkaline phosphatase > 2.5 times ULN
  * Uncontrolled hypercalcemia (defined as serum calcium > 14 mg/dL)
  * Serum creatinine > 2.0 mg/dL or creatinine clearance of < 30 mL/min
  * ANC < 1000 cells/mm3 or < 750 cells/mm3 due to >50% marrow involvement
  * Platelet count < 50,000 cells/mm3
  * Hemoglobin < 8.0 g/dL
* Patient is known to be human immunodeficiency virus (HIV)-positive.
* Patient is known to be hepatitis B surface antigen-positive or has known active hepatitis C infection.
* Patient has an active systemic infection requiring treatment or within 14 days before first dose of PRLX 93936.
* Pregnant or nursing women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-03; Primary Completion 2014-03 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | Cycle 1 (28 days from first dose)

SECONDARY OUTCOMES:
Response to treatment | Each cycle (assessed every 28 days starting from first dose, for up to 8 months)
Time to response | From date of first dose to date of response, assessed up to 8 months
Duration of response | From date of response to first documented progression or death, or date last known progression-free and alive at study discontinuation, assessed up to 8 months
Time to progression | From date of first dose to first documented progression, assessed up to 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Paul Richardson, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (6):
- United States (6):
  - Tufts Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Sarah Cannon Research Institute, Nashville, Tennessee